CLINICAL TRIAL: NCT06704373
Title: Effect of Thoracic Manipulation on Peripheral Muscle Oxygenation, Pain, and Disability in Office Workers With Back Pain
Brief Title: The Effects of Thoracic Manipulation on Peripheral Muscle Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alev-Man24
Record Dates: First submitted 2024-10-02; First posted 2024-11-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Back Pain; Spine Stiffness; Sedentary Behavior; Disability Physical
Keywords: moxy; spinal pain; sedantary; chiropractic
MeSH Terms: conditions — Back Pain; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into intervention (manipulation group) and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manipulation group (Experimental): Thoracic spinal manipulation will be performed between the T1-T12 vertebral levels, based on the segment with movement limitations. The manipulation will be applied to the area of back pain using a high-velocity, low-amplitude thrust with a short-lever technique.
  Also, the same postural exercises that were given to the control group will be given.
  Interventions: Other: thoracal manipulation; Other: Exercise
- Control Group (Active Comparator): The postural exercises program will be given.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: thoracal manipulation — Thoracal manipulation will be applied only one session.
  Arms: Manipulation group
Other: Exercise — Both groups will perform the same postural exercises, which will be applied twice a week for 4 weeks. The intervention group will receive thoracic manipulation for one session.
  Other Names: Postural Exercise

SUMMARY:
Office workers spend 70-85% of their time sitting, which leads to postural disorders and musculoskeletal system diseases. Back pain is the most common health problem among office workers who need to sit. Studies have shown that spinal manipulation can help reduce back pain by decreasing the stiffness of spine segments associated with joint dysfunction. The primary aim of this study is to investigate the effects of thoracic spinal manipulation on peripheral oxygenation, pain, and disability of the back muscles in office workers with back pain, at acute, 10-day, and 4-week follow-up periods. The secondary aim is to evaluate whether the parameters have a significant relationship.

The study will include volunteers aged 20-50 who are active office workers with no orthopedic, neurological, or psychological disorders, who have experienced back pain in the last 3 months, and who have a numerical pain scale score of at least 30 mm out of 100 mm. Participants will be randomized into the thoracic spinal manipulation and the control groups. Both groups will receive postural exercises. The thoracic spinal manipulation group will receive a single session of spinal manipulation, while the control group will only receive postural exercises. The study is expected to find significant improvement in peripheral muscle oxygenation, back pain, and disability scores following thoracic spinal manipulation. This study aims to contribute to the literature by focusing on how peripheral muscle oxygenation is affected by thoracic spinal manipulation.

DETAILED DESCRIPTION:
Office workers spend 70-85% of their time sitting at their workplaces, with an average working time of 8 hours. This prolonged inactivity can lead to serious health issues such as musculoskeletal disorders, repetitive movements, static postures, and improper body positions. Due to their limited mobility, office workers are at risk of experiencing problems with their body postures. Studies have shown that back pain is a common issue among office workers. However, thoracic spine pain between the T1-T12 vertebrae is less studied and less debilitating than cervical and lumbar pain. The most common causes of back pain are muscle tension, trauma, acute injury, strain, or poor posture. The posture, mobility, and stability of the thoracic spine are important factors in pain syndromes and degenerative changes. The success of treatment relies on understanding the anatomy and biomechanics of the spine. Research on mechanoreceptor effects is significant for manual therapy, including spinal manipulation and mobilization techniques. These therapies target intervertebral joints and affect adjacent joints and surrounding soft tissues. Chiropractic spinal manipulation, performed by professionals at the intersection of traditional and alternative medicine, has been found effective in treating back pain and reducing pain. Thoracic spinal manipulation may help relax spinal segments associated with secondary muscle spasms due to joint dysfunction. Studies have shown significant improvements in range of motion and pain in the acute period following thoracic manipulation. Spinal manipulation combined with exercise can enhance an individual's quality of life and improve pain conditions.

NIRS (near-infrared spectroscopy) has been used to measure the oxygen status of muscle tissue, demonstrating the balance between muscle oxygen delivery and tissue V̇O2. The fascial system encompassing the large muscle groups in the back can lead to muscle overload, reducing blood flow and creating myofascial adhesions. A recent study presented initial evidence that myofascial reorganization techniques could improve trapezius muscle tissue oxygenation and peripheral blood flow in patients with neck pain.

To our knowledge, there are no studies evaluating the effect of spinal manipulation on muscle oxygenation in individuals with back pain. Our research aims to contribute to the literature by examining the changes in oxygenation, pain, and disability in the upper trapezius and interscapular region and lumbar spine muscles following a single session of thoracic spinal manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Active desk-based office worker for the past 3 months
* Age between 20 and 50 years
* Back pain experience in the last 3 months
* Willing to participate in the study

Exclusion Criteria:

* Diagnosis of osteoporosis
* Presence of a newly formed fracture
* Recent trauma
* Cancer
* Osteomyelitis
* Hypermobility
* Ankylosing spondylitis
* Presence of an aneurysm
* Presence of vascular occlusion
* Malignancies

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Periferal muscle oxygen measurement | Baseline, right after intervention, ten days after post intervention, four weeks after post intervention
  Muscle oxygen levels will be measured using the Moxy Monitor. The Moxy Monitor is a mobile, non-invasive method for measuring SmO2. The device uses near-infrared spectroscopy (NIRS) technology and features a patented algorithm that measures hemoglobin and myoglobin in capillaries and muscle tissues with a wearable monitor. Moxy device measures real-time muscle oxygenation (SmO2) and total hemoglobin (tHb) levels by using near-infrared spectroscopy.

SECONDARY OUTCOMES:
Oswestry Disability Index | Baseline, right after intervention, ten days after post intervention, four weeks after post intervention
  The survey consists of ten items related to pain severity, sitting, standing, and social life, with each item rated by participants on a scale from 0 to 5. The total score is calculated by dividing the patient's score by the possible maximum score and then multiplying by 100. Therefore, the score of the Oswestry Disability Questionnaire ranges from 0 to 100, with a higher score indicating greater disability.
Neck Disability Index | Baseline, right after intervention, ten days after post intervention, four weeks after post intervention
  The Neck Disability Index (NDI) comprises ten items that assess the impact of neck pain on daily activities, including personal care, lifting, reading, and social life. Each item is rated by participants on a scale from 0 to 5, with higher scores indicating greater disability. The total score is calculated by dividing the participant's score by the maximum possible score and then multiplying by 100. Consequently, the NDI score ranges from 0 to 100, where a higher score reflects a higher level of disability associated with neck pain.
Numeric Pain Scale | Baseline, right after intervention, ten days after post intervention, four weeks after post intervention
  The Numeric Pain Scale (NPS) is a subjective measure used to assess pain intensity, where participants rate their pain on a scale from 0 to 100 mm. A score of 0 indicates no pain, while a score of 100 represents the worst imaginable pain. Participants mark their pain level on a line, and the distance from the zero point is measured to obtain the score.

CONTACTS AND LOCATIONS:
Overall Officials: Alev Atasever, PT, Principal Investigator — Bahcesehir University, Graduate Education Institute,Chiropractic Master of Science Program; Pelin Pişirici, PT, PhD, Study Director — Bahcesehir University, Faculty of Health Sciences; Berkay Eren Pejlivanoğlu, PT, PhD, Study Chair — Bahcesehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation
Locations (1):
- Bahcesehir University, Beşiktaş, Istanbul, Turkey (Türkiye)